CLINICAL TRIAL: NCT07069413
Title: Sibwatch: Optimizing Intervention Options for Infants and Toddlers With a High Likelihood of Social Communication Delays and Language Disorder
Brief Title: Sibwatch: Optimizing Intervention Options for Infants and Toddler Siblings of Autistic Children
Acronym: Sibwatch
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Lauren Hampton, Assistant Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY00006726
Record Dates: First submitted 2025-06-30; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-06

CONDITIONS: Autism Sibling
Keywords: autism
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: All outcomes assessment ratings will be conducted by an assessor naive to treatment condition. All assessments will be administered by an assessor also naive to treatment condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Business as Usual (No Intervention): Control arm where participants will receive community treatments, as usual.
- tele-ImPACT (Experimental): Participants will receive 12 weeks of intervention
  Interventions: Behavioral: tele-ImPACT

INTERVENTIONS:
Behavioral: tele-ImPACT — Participants will receive 12 weeks of Project ImPACT intervention as delivered via Telehealth
  Arms: tele-ImPACT

SUMMARY:
This rigorous randomized controlled trial will evaluate the efficacy and acceptability of a preemptive, telehealth intervention (tele-ImPACT) in a large, representative sample of infant siblings of autistic children, who are known to be at high likelihood of receiving a future diagnosis of autism and/or developmental language disorder (HL-Sibs). If our hypotheses are supported, this innovative and interdisciplinary study will provide empirical support for a novel approach to treatment that is theoretically motivated and developmentally informed, as well as accessible for and acceptable to families, and will lend new insights into the developmental windows in which, mechanisms by which, and subgroups for which the treatment works. Such findings would have strong implications for research, policy, theory, and practice in young children at risk for autism and/or language disorder.

DETAILED DESCRIPTION:
Autism is a neurodevelopmental condition that is highly prevalent and that comes at a high cost to affected children and their families. The costs of autism can be attributed, at least in part, to the effects of the condition on children's social communication and language development. Younger siblings of autistic children (HL-Sibs) are highly likely to receive a future diagnosis of autism and/or language disorder themselves. Even those HL-Sibs who are not diagnosed have an increased likelihood of displaying differences in social communication and delays in language development. There is increasing support that preemptive interventions may influence caregivers' use of strategies that scaffold development and translate to effects on social communication and language skills in HL-Sibs. However, prior studies of preemptive interventions have been limited by the inclusion of samples that are rather homogenous, likely reflecting those families who can readily access the medical centers and academic institutions conducting this research. Additionally, past investigations suggest that effects of preemptive interventions may (a) yield only indirect effects on child social communication and language, and (b) vary according to child and caregiver factors, but no previously identified mediators or moderators of preemptive intervention effects have been replicated, and many factors that likely explain or influence differential intervention effects have not yet been explored. Further, the extant literature testing the efficacy of preemptive interventions has administered treatments across a broad range of child ages, and researchers do not yet know precisely when preemptive treatment is most likely to yield favorable effects. Finally, some studies have reported high rates of attrition amongst families assigned to treatment, suggesting that caregivers may not find preemptive interventions to be acceptable. The present study will, thus, evaluate the efficacy of ImPACT, an intervention that is established for use with autistic children and that has amassed some past empirical support as delivered in vivo in HL-Sibs, as administered by telehealth (hereafter referred to as tele-ImPACT) relative to a no-treatment control for effects on caregiver strategy use, proximal child skills, and distal child social communication and language in a large, representative sample in the context of a rigorous randomized clinical trial. Advanced analytic approaches will be employed to test numerous putative moderators and mediators of tele-ImPACT effects, and qualitative approaches will be utilized to assess the acceptability of the candidate treatment amongst caregivers. INNOVATION AND IMPACT: This innovative and interdisciplinary study is expected to (a) provide empirical support for a novel preemptive intervention that is theoretically motivated and developmentally informed, as well as accessible for and acceptable to families affected by autism in the United States, and (b) lend new insights into the developmental windows in which, mechanisms by which, and the subgroups for which this intervention works. Such findings would have strong implications for theory, policy, research, and clinical practice in young children at elevated likelihood for autism and developmental language disorder.

ELIGIBILITY:
Inclusion Criteria:

* chronological age between 6-24 months
* has at least one older biological sibling diagnosed with autism

Exclusion Criteria:

* adverse neurological history
* primary sensory deficit (hearing or visual impairment)
* pre-term birth (gestation <37 weeks)
* pre-existing diagnosis of autism or language delay

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2031-03-31 (Estimated); Study Completion 2032-03-31 (Estimated)

PRIMARY OUTCOMES:
Child Social Communication | 9 months
  A single z-score average of two scales: VABS socialization standard score and ADOS-2 reflected social affect calibrated severity score
Child Receptive Language | 9 months
  A single z-score average of two scales: MSEL receptive scaled score and VABS expressive scaled score
Child Expressive Language | 9 months
  A single z-score average of two scales:MSEL expressive scaled score, VABS expressive scaled score

IPD SHARING:
Plan to Share IPD: Undecided